CLINICAL TRIAL: NCT00150566
Title: A Phase IIIb, Multi-center, Two-Cohort, Randomized Study, With an Open-Label Run-In and a Long-Term Extensions Phase, Assessing an Extended Dose Range of Lanthanum Carbonate in End Stage Renal Disease Subjects Receiving Hemodialysis
Brief Title: Efficacy and Safety of Lanthanum in Controlling Serum Phosphate Levels in Subjects With End Stage Renal Disease Who Require Treatment for High Levels of Phosphate in Their Blood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD405-312
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate

SUMMARY:
The purpose of this study is to test how well higher doses of lanthanum carbonate reduce the pre-dialysis level of serum phosphorus in subjects undergoing dialysis due to end stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ESRD who currently require treatment for hyperphosphatemia
* Women of childbearing potential must have a negative serum beta HCG pregnancy test and must agree to abstain from sexual activity or to use acceptable contraceptives from the time of informed consent throughout the study

Exclusion Criteria:

* Treatment with compounds containing calcium, aluminum or magnesium for use as a phosphate binder
* Hypocalcaemia
* Treatment-naive to any phosphate binder with a serum phosphorus < 5.5 mg/dL
* Any significant gastrointestinal surgery or gastrointestinal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460
Dates: Start 2004-02-09 (Actual); Primary Completion 2005-10-08 (Actual); Study Completion 2005-10-08 (Actual)

PRIMARY OUTCOMES:
Pre-dialysis serum phosphate levels after 4 and 8 weeks of treatment | 4 & 8 weeks

SECONDARY OUTCOMES:
Tolerability | 8 weeks
Quality of Life | 8 weeks
Subject/physician satisfaction and preference questionnaires | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Mehrotra R, Martin KJ, Fishbane S, Sprague SM, Zeig S, Anger M; Fosrenol Overview Research Evaluation Study for Early Experience Study Group. Higher strength lanthanum carbonate provides serum phosphorus control with a low tablet burden and is preferred by patients and physicians: a multicenter study. Clin J Am Soc Nephrol. 2008 Sep;3(5):1437-45. doi: 10.2215/CJN.04741107. Epub 2008 Jun 25. PMID 18579668
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html